CLINICAL TRIAL: NCT01188356
Title: AssEssment of CoMorbidities & Atrial ArRhythmiA Burden in DuaL-Chamber PaceD Patients
Brief Title: EMERALD - AssEssment of CoMorbidities & Atrial ArRhythmiA Burden in DuaL-Chamber PaceD Patients
Acronym: EMERALD
Status: Completed | Type: Observational
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Other Study IDs: RGST04-EMERALD Study; RGST04
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Atrial Arrhythmia
Keywords: Reply; Symphony; Atrial arrhythmias; V pacing; Evaluate the incidence and evolution over-time of co-morbidities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the incidence and evolution over-time of co-morbidities in a general dual-chamber pacemaker population (n=2188 patients) through a 2 years follow-up.

DETAILED DESCRIPTION:
The study will focus on the number of patients moving to persistent Atrial Fibrillation as a function of cumulative %Vp (< or >40%), in a general dual-chamber pacemaker population through a 2 year follow-up (n=2188).

The same endpoint will be analyzed in sub populations (Sinus Node Disease and AVB) at 4 years follow up (n=4290).

ELIGIBILITY:
Inclusion Criteria:

- Patient implanted (primo-implant, replacement, upgrade) with dual chamber pacemaker from less than two months or implanted at inclusion.

Exclusion Criteria:

* Contraindicated for cardiac pacing, according to the ESC and ACC/AHA/HRS guidelines
* Permanent or persistent atrial tachyarrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sponsor plans the enrolment of a total of 2188 subjects in this clinical investigation.
Sampling Method: Probability Sample
Enrollment: 4350 (Actual)
Dates: Start 2010-03; Primary Completion 2015-04 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Atrial arrhythmias incidence | 2 years
  Two consecutive visits in which atrial fibrillation was present or - at least 22 hours of atrial fibrillation for at least 7 consecutive days or - at least 22 hours of atrial fibrillation per day for fewer than 7 consecutive days if an interruption by electrical or pharmacologic cardioversion occurred
% ventricular pacing | 2 years
  as measured in the device over the timeframe period

CONTACTS AND LOCATIONS:
Locations (190):
- United States (32):
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Mountain Vista Medical Center, Mesa, Arizona
  - Pacific Arrhythmia Services, Mesa, Arizona
  - Peoria, Arizona
  - Advanced Heart and Vascular Institute, Phoenix, Arizona
  - Harishchandra N. Patel, M.D., Inc., Anaheim, California
  - Narayan R. Devaraj, M.D., Inc., Anaheim, California
  - St. Rose Hospital, Fremont, California
  - Hanford, California
  - Los Angeles, California
  - Simi Valley Hospital, Simi Valley, California
  - Metroform Medical Complex, Newark, Delaware
  - Complete Cardiology Care Live Oak Street, New Smyrna Beach, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cardiology, Atlanta, Georgia
  - Northeast Georgia heart Center, Gainesville, Georgia
  - Electrophysiology Research Foundation, Warren Township, New Jersey
  - Abbas Shehadeh, MD, PA, West Orange, New Jersey
  - Low Country Medical Group, Beaufort, North Carolina
  - Charlotte, North Carolina
  - East Ohio Rag Hospital, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Toledo Clinic Inc, Toledo, Ohio
  - Lakshimi Mizin Cardiology, Carbondale, Pennsylvania
  - Scranton Heart Institute, Clarks Green, Pennsylvania
  - Easton Cardiology, Easton, Pennsylvania
  - Coastal Cardiology, Charleston, South Carolina
  - Charleston, South Carolina
  - Columbia Cardiology Consultants, Columbia, South Carolina
  - Ocean Cardiology, Murrells Inlet, South Carolina
  - Pawleys Island, South Carolina
  - Victoria Heart and Vascular Center, Victoria, Texas
- John Flynn Private Hospital, Tugun, Queensland, Australia
- Belgium (8):
  - Cliniques Sud Luxembourg, Arlon
  - RHMS Ath - Baudour, Baudour
  - Hôpital Brugmann, Brussels
  - vzw Sint-Jozefskliniek, Izegem
  - AZ Groeninge, Kortrijk
  - UZ Gasthuisberg Leuven, Leuven
  - Clinique & Maternité Sainte-Elisabeth Namur, Namur
  - Hôpital de La Tourelle, Verviers
- Canada (4):
  - Hotel Dieu de Montreal, Montreal
  - Maisonneuve-Rosemont, Montreal
  - Chus-Fleurimont - Hospital, Sherbrooke
  - Trois-Rivières
- Denmark (2):
  - Bispebjerg Hospital, Bispebjerg
  - Gentofte Hospital, Hellerup
- France (50):
  - Polyclinique Parc Rambot, Aix-en-Provence
  - CHG Albi, Albi
  - Centre hospitalier de la Région d'Annecy, Annecy
  - Cabinet médical, Arras
  - Chu Brest, Brest
  - CH Brive, Brive-la-Gaillarde
  - Clinique Ste Marie, Cambrai
  - Ch Chaumont, Chaumont
  - CH Châlon en Champagne, Châlon-en-Champagne
  - Clinique Bon Secours, Châtellerault
  - Ch Cherbourg, Cherbourg
  - HIA Percy, Clamart
  - CH René Pleven, Dinan
  - CH Douarnenez, Douarnenez
  - Centre Cardiologique d'Evecquemont, Évecquemont
  - CH D'Evreux, Évreux
  - CMCO, Évry
  - CH de Firminy, Firminy
  - Hagondange
  - CH de la région St Omer, Helfaut
  - Cabinet de cardiologie, Hénin-Beaumont
  - Cabinet de cardiologie, Lannion
  - Centre Hospitalier Pierre Le Damany, Lannion
  - Cmc Parly Ii, Le Chesnay
  - CH J. Monod, Le Havre
  - CH St Philibert, Lomme
  - CH de Bretagne Sud, Lorient
  - Ch de Bretagne Sud, Lorient
  - Centre Hospitalier de Sambre Avesnois, Maubeuge
  - Hôpital Ste Blandine, Metz
  - Clinique Claude Bernard, Metz
  - Clinique de Montargis, Montargis
  - Clinique Pont de Chaume, Montauban
  - Cabinet de Cardiologie, Narbonne
  - Hopital Privé A. Brillard, Nogent-sur-Marne
  - Hôpital Lariboisière, Paris
  - CH Poitiers, Poitiers
  - Centre hospitalier général, Roanne
  - Clinique Saint Hilaire, Rouen
  - Centre hospitalier Yves Le Fol, Saint-Brieuc
  - CCN, Saint-Denis
  - CHU - Hôpital Nord, Saint-Etienne
  - H.I.A. Begin, Saint-Mandé
  - CHG, Saint-Nazaire
  - CH, Soissons
  - CH Broussais, St-Malo
  - Centre Hospitalier, Tulle
  - Centre Hospitalier de Valence, Valence
  - Ch Valenciennes, Valenciennes
  - CH Vannes - CH Bretagne Atlantique, Vannes
- Germany (47):
  - Kardiologische Praxis Dr. Schröter, Alten
  - PRAXIS, Annaberg-Buchholz
  - Praxis Dr. Gerhard BÖHM, Arnstadt
  - Dr. med. Kai-Uwe Westermann, Aschersleben
  - FOWIS e. V., Förderverein für die medizinische Wissenschaft und Schulung, Berlin
  - Praxis Dr. Bott, Berlin
  - Praxis Schmidt/Engelsing, Berlin
  - Berlin
  - Innere Medizin und Kardiologie, Bünde
  - Praxis Dr. Gloes, Chemnitz
  - Praxis Dr. Med Stellmach, Chemnitz
  - Praxis Troeger, Chemnitz
  - Gesundheitszentrum Im Esc, Dresden
  - Praxis Engelhard Kaiser, Düsseldorf
  - Kardiologische Praxis, Ebersbach
  - FA fur Innere Medizin/Kardiologie, Eilenburg
  - Klinik Eilenburg, Eilenburg
  - Kardiologische Praxis, Eschwege
  - Gemeinschaftspraxis Dr. Bemmann, Dr. Sadowski, Dr. Boehme, Frankfurt
  - Kardiocentrum Frankfurt and der Klinik Rotes Kreuz, Frankfurt
  - DRK Krankenhaus Grevesmuehlen, Grevesmühlen
  - Baerenfaenger Dr. Petra Private Practice, Hanau
  - Gemeinschaftspraxis Dr. Loebe - Dr. Weissbrodt, Leipzig
  - FA fur Innere Medizin/Kardiologie, Leipzig
  - Praxis Dr. Andreas Herzfeld, Leipzig
  - Praxis Dr. med. Irina Boran, Leipzig
  - Praxis Schreiner, Leipzig
  - Medizin/Kardiologie/Diabetologie, Lichtentanne
  - Staedt. Linikum Medizinische Klinik Lueneburg, Lüneburg
  - SPENGLER, Machern
  - PRAXIS, Markkleeberg
  - Memmingen
  - Kardiologische - angiologische Praxis Dr. med. Jörg Walter, Mühlhausen
  - Klinikum Bogenhausen, München
  - Gemeinschaftspraxis Dres.Med.U. Heinrich Und Dr Predel, Nordhausen
  - Praxis für Gefäßmedizin, Nordhausen
  - Praxis Dr. Donaubauer, Oschatz
  - Praxis Dr. Stuehn-Pfeiffer , Dr. Wilke, Papenburg
  - Med. Martina Trummel Praxis Innere Medizin / Kardiologie, Quedlinburg
  - DRK Krankenhaus Ratzeburg, Ratzeburg
  - Praxis Dr. Noehring, Schwarzenberg
  - Diakonie Klinikum Schwäbisch Hall GmbH, Schwäbisch Hall
  - Praxis Prof. Frey, Starnberg
  - Praxis Dr. Birkenhagen, Stollberg
  - Sohien und Hufeland Klinikum Weimar Gmbh, Weimar
  - Praxis Dr Lebek, Wunsiedel
  - Praxis Dr. Brode, Zwickau
- Italy (10):
  - Ospedale San Donato, Arezzo
  - Ospedale Civile di Conegliano, Conegliano
  - Arcispedale S. Maria Nuova, Florence
  - Ospedale Nuovo San Giovanni di Dio, Florence
  - Ospedale S. Maria Annunziata, Florence
  - AOU S.Paolo, Milan
  - Ospedale Valdarno, Montevarchi
  - Ospedale Sacrocuore - Don Calabria, Negrar
  - University Hospital of Pisa, Pisa
  - Ospedale OO.OO.San Giovanni e Ruggi d'Aragona, Salerno
- Japan (12):
  - Shobara Red Cross Hospital, Hiroshima
  - Kimitsu Chuo Hospital, Kisarazu
  - Yokosuka Kyosai General Hospital, Kyosai
  - Sakurabashi Watanabe Hospital, Osaka
  - Tominaga Hospital, Osaka
  - Osaka National Hospital, Osaka
  - National Hospital Organization Oita Medical Center, Ōita
  - Okamura Memorial Hospital, Suntou-gun
  - Tokai University Tokyo Hospital, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Tokyo
  - Aoyama Hospital, Toyokawa
  - Yokohama City University Hospital, Yokohama
- Gelre Ziekenhuizen, Zutphen, Netherlands
- Spain (19):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Marina Salud de Denia, Denia
  - Hospital general de Elda, Elda
  - H.A. Marcide, Ferrol
  - Hospital Galdakao, Galdakao
  - Cabuenes, Gijón
  - Hospital Universitario San Cecilio, Granada
  - Hospital Rafael Mendez, Lorca
  - Complejo Hospitalario Xeral Calde, Lugo
  - Hospital 12 de Octubre, Madrid
  - Hospital de Fuenlabrada, Madrid
  - CHOU, Ourense
  - Hospital Montecelo, Pontevedra
  - Virgen del Rocio, Seville
  - Joan XXIII, Tarragona
  - Hospital Clínico Universitario, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Lluis Alcanyis, Xàtiva
- Switzerland (4):
  - Basel
  - Lausanne
  - Ospedale La Carità, Locarno
  - Universitaetsspital Zuerich, Zurich